CLINICAL TRIAL: NCT04466280
Title: Efficacy and Safety of Mucoadhesive Sustained Release, Mucodentol, in Comparison With Hydroxychloroquine to Prevent COVID-19 Disease in Healthcare Providers at Baqiyatallah Hospital in Tehran
Brief Title: Efficacy and Safety of Mucoadhesive Sustained Release, Mucodentol, in Comparison With Hydroxychloroquine to Prevent COVID-19
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The financier of this research project died due to covid-19, Therefore, this project was stopped due to lack of funds
Sponsor: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Principal Investigator, Mohammad Sadegh Bagheri Baghdasht, Principal Investigator, Baqiyatallah Medical Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IR.BMSU.REC.1399.086
Record Dates: First submitted 2020-07-09; First posted 2020-07-10 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Personal Protective Equipment

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): Participants in this group use personal protective equipment in the face of patients with COVID-19
  Interventions: Device: Personal protective equipment
- Intervention Group 1 (Experimental): In this group, participants will receive 200 mg of hydroxychloroquine tablets daily in addition to personal protective equipment.
  Interventions: Drug: Hydroxychloroquine; Device: Personal protective equipment
- Intervention Group 2 (Experimental): In this group, participants, while observing and using complete personal protective equipment, will apply a thin layer of Dentol gel to the vestibular area of the mouth daily, every 6 to 8 hours.
  Interventions: Drug: Mucodentol; Device: Personal protective equipment

INTERVENTIONS:
Drug: Hydroxychloroquine — 200 mg of hydroxychloroquine daily for participants in the intervention group 1
  Arms: Intervention Group 1
Drug: Mucodentol — Intervention Group 2 participants will place a thin layer of Dentol gel in the vestibular area of the mouth every 6 to 8 hours.
  Other Names: Dentol Gel
  Arms: Intervention Group 2
Device: Personal protective equipment — Personal protective equipment such as masks, gloves, protective shields

SUMMARY:
180 people from the medical staff and high-risk people in Baqiyatallah Hospital, who are in close contact with patients, will enter the study. Participants will be divided into two intervention groups and one control group. The control group will use the full protective equipment assigned to the treatment staff. In addition to protective equipment, the first intervention team will receive a daily diet of 200 mg hydroxychloroquine tablets. The second intervention team, while observing and using the complete protective equipment, will place a thin layer of Mucodentol gel in the vestibular area of the mouth daily, every 6 to 8 hours.

At the beginning of the treatment, qualified people will participate in the study while recording demographic and clinical information, PCR test will be performed, and if they have negative PCR, they will be in one of the 3 study groups. During the study, if the symptoms of the disease occur in each of the participants, the test will be taken again. If the test is positive, the person will withdraw from the study, and the patient's information will be recorded. Finally, the people present in the study will be tested for PCR, and the results of the disease and the side effects of the drugs will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Negative PCR testing through throat swabs
* Signing Conscious Consent

Exclusion Criteria:

* History of ocular complications and visual disturbances
* Sensitivity to plant compounds in the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
PCR test | up to 1 month
  Laboratory PCR testing can help diagnose the disease

SECONDARY OUTCOMES:
Laboratory Treatment Response | up to 1 month
  Normal blood cell count and CRP count (normal laboratory range)
drug reactions Adverse | up to 1 month
  Complications in both groups should be evaluated and evaluated during treatment.
Allergic drug | up to 1 month
  There will be known allergic reactions to the drugs.
Radiological Treatment Response | up to 1 month
  CT scans help determine how much the lungs are affected by COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Sadegh Bagheri Baghdasht, Tehran, Iran